CLINICAL TRIAL: NCT04011865
Title: Robot-assisted vs Laparoscopic Radical Prostatectomy for Prostate Cancer Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Binh Dan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BD022019
Record Dates: First submitted 2019-05-13; First posted 2019-07-09 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer
Keywords: laparoscopic radical prostatectomy; robotic-assisted laparoscopic radical prostatectomy; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic-assisted surgery (Active Comparator)
  Interventions: Procedure: Radical prostatectomy
- Laparoscopic surgery (Sham Comparator)
  Interventions: Procedure: Radical prostatectomy

INTERVENTIONS:
Procedure: Radical prostatectomy — The patients diagnosed with prostate cancer (local or locally advanced stages) will be allocated to the study for performing radical prostatectomy surgery.

SUMMARY:
This study is to compare the outcomes of robotic-assisted laparoscopic radical prostatectomy (RARP) and laparoscopic radical prostatectomy (LRP) for prostate cancer treatment in terms of perioperative surgical, functional and oncological outcomes.

DETAILED DESCRIPTION:
Participants will either have robotic-assisted laparoscopic radical prostatectomy (RARP) or laparoscopic radical prostatectomy (LRP) as determined by the treating surgeon. All participants will undergo tests and questionnaires to determine urinary and erectile function, biopsies to determine perioperative surgical, functional and oncological outcomes. These assessments will be conducted pre-operatively, post-operatively and at certain follow-up time points up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men aged 18 years and over;
2. Undergoing RARP or LRP. prostatectomy for prostate cancer at Binh Dan Hospital;
3. Clinically suitable for radical prostatectomy (cT1-3, No, Mo);
4. Cognitively able to give written informed consent for participation;
5. Elective procedure.

Exclusion Criteria:

1. The patient lacks the ability to consent for themselves;
2. Patients unwilling to undergo pre- and post-operative evaluation according to the protocol;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The console time | During the surgery
  The time which surgeon spends on the robot console by minuite
Mean of blood loss | During the surgery
  Milliliter
Perioperative transfusion rate (%) | Up to 1 month after operation
  The number of cases which will be transfused.
The rate of positive surgical margins, extracapsular extension, seminal vesicle invasion, (5)perineural invasion, the number of lymph node yield and node involvement, | Up to 1 week after operation
  Number of cases, based on the result of pathology.
Number of blood units transfused | Up to 1 week after operation
  Milliliter
the rate of conversion to open surgery, the rate of intraoperative incidents (%), | Up to 1 weeks after the surgery.
  Percentage
The postoperative recovery parameters using Numeric Pain Rating Scale (NPRS), | Up to 3 month after surgery
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of pain, in a total of 10 points, higher score means worse, with 0 means no pain and 10 is the worst pain. The mean score will be calculated to reflect the post-operative pain.
Change of hemoglobin from baseline | Up to 1 week after operation
  (mg/mL)
The drainage time | Up to 3 months after surgery
  (day),
To assess urethral catheter time, urethral catheter time | Up to 3 months after surgery
  (day)
To assess bowel movement recovery time, | Up to 1 week after surgery
  (day)
To assess postoperative hospital stay | Up to 1 month after surgery
  (day)
The rate of postoperative complications (including infections) | in day 3, day 7, and 1 month after surgery.
  Percentage
PSA level in blood | Before operation
  (mg/mL)
PSA level in blood | 6 weeks post-operation
  (mg/mL)
PSA level in blood | 3 months post-operation
  (mg/mL)
PSA level in blood | 6 months post-operation
  (mg/mL)
PSA level in blood | 12 months post-operation
  (mg/mL)
local and regional recurrences on sonography | through study completion, an average of 1 year
  including ultrasound when PSA rising or any indication of recurrent
local and regional recurrences, on MRI | through study completion, an average of 1 year
  including MRI when PSA rising or any indication of recurrent
local and regional recurrences, on PET Scan | through study completion, an average of 1 year
  including PET Scan, when PSA rising or any indication of recurrent

SECONDARY OUTCOMES:
Evaluating the pre and postoperative lower urinary tract symptoms using Full score of International Prostate Symptoms Scores (IPSS) | Preoperative
  It contains seven questions related to symptoms related to BPH and one question related to the patient's perceived quality of life. The symptoms must have been experienced in the last month and each answer is scored from 0 to 5 for a maximum score of 35 points. The sum score will be calculated and the mean score will be evaluated.
Evaluating the pre and postoperative lower urinary tract symptoms using International Prostate Symptoms Scores (IPSS) | 3 months postoperative
  It contains seven questions related to symptoms related to BPH and one question related to the patient's perceived quality of life. The symptoms must have been experienced in the last month and each answer is scored from 0 to 5 for a maximum score of 35 points. The sum score will be calculated and the mean score will be evaluated.
Evaluating the pre and postoperative lower urinary tract symptoms using Full score of International Prostate Symptoms Scores (IPSS) | 6 months, postoperative
  It contains seven questions related to symptoms related to BPH and one question related to the patient's perceived quality of life. The symptoms must have been experienced in the last month and each answer is scored from 0 to 5 for a maximum score of 35 points. The sum score will be calculated and the mean score will be evaluated.
Evaluating the pre and postoperative lower urinary tract symptoms using Full score of International Prostate Symptoms Scores (IPSS) | 12 months postoperative.
  It contains seven questions related to symptoms related to BPH and one question related to the patient's perceived quality of life. The symptoms must have been experienced in the last month and each answer is scored from 0 to 5 for a maximum score of 35 points. The sum score will be calculated and the mean score will be evaluated.
Erectile function assessments questionnaires and scoring using Index of Erectile Function Questionnaire, IIEF5, full score | Preoperative
  The 15-question International Index of Erectile Function (IIEF) Questionnaire is a validated, multi-dimensional, self-administered investigation that has been found useful in the clinical assessment of erectile dysfunction and treatment outcomes in clinical trials. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction. The score ranges from 22 - 25 for Normal erectile function (no ED), 17 - 21 for Mild ED, 12 - 16 for Mild to moderate ED, 8 - 11 for Moderate ED, and from 1 - 7 for Severe ED (5 - 7, if a man had no opportunity to engage in sexual activity). The mean score will be calculated.
Erectile function assessments questionnaires and scoring using Index of Erectile Function Questionnaire, IIEF5, full score | 3 months, postoperative
  The 15-question International Index of Erectile Function (IIEF) Questionnaire is a validated, multi-dimensional, self-administered investigation that has been found useful in the clinical assessment of erectile dysfunction and treatment outcomes in clinical trials. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction. The score ranges from 22 - 25 for Normal erectile function (no ED), 17 - 21 for Mild ED, 12 - 16 for Mild to moderate ED, 8 - 11 for Moderate ED, and from 1 - 7 for Severe ED (5 - 7, if a man had no opportunity to engage in sexual activity). The mean score will be calculated.
Erectile function assessments questionnaires and scoring using Index of Erectile Function Questionnaire, IIEF5, full score | 6 months, postoperative.
  The 15-question International Index of Erectile Function (IIEF) Questionnaire is a validated, multi-dimensional, self-administered investigation that has been found useful in the clinical assessment of erectile dysfunction and treatment outcomes in clinical trials. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction. The score ranges from 22 - 25 for Normal erectile function (no ED), 17 - 21 for Mild ED, 12 - 16 for Mild to moderate ED, 8 - 11 for Moderate ED, and from 1 - 7 for Severe ED (5 - 7, if a man had no opportunity to engage in sexual activity). The mean score will be calculated.
Erectile function assessments questionnaires and scoring using Index of Erectile Function Questionnaire, IIEF5, full score | 12 months postoperative
  The 15-question International Index of Erectile Function (IIEF) Questionnaire is a validated, multi-dimensional, self-administered investigation that has been found useful in the clinical assessment of erectile dysfunction and treatment outcomes in clinical trials. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction. The score ranges from 22 - 25 for Normal erectile function (no ED), 17 - 21 for Mild ED, 12 - 16 for Mild to moderate ED, 8 - 11 for Moderate ED, and from 1 - 7 for Severe ED (5 - 7, if a man had no opportunity to engage in sexual activity). The mean score will be calculated.
The quality of life questionnaires and scoring using the the Short Form (36) Health Survey questionnaire | Preoperative
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. The mean score will be calculated.
The quality of life questionnaires and scoring using the the Short Form (36) Health Survey questionnaire | 3 months, postoperative.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. The mean score will be calculated.
The quality of life questionnaires and scoring using the the Short Form (36) Health Survey questionnaire | 6 months, postoperative
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. The mean score will be calculated.
The quality of life questionnaires and scoring using the the Short Form (36) Health Survey questionnaire | 12 months postoperative
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. The mean score will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Hung V Tran, MD, PhD, Study Director — Binh Dan Hospital
Locations (1):
- Binh Dan Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No